CLINICAL TRIAL: NCT00842062
Title: Study of the MyoScience Tissue Remodeling Device for Facial Rejuvenation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-3000
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Facial Rhytides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MyoScience Tissue Remodeling Device (Experimental)
  Interventions: Device: MyoScience Tissue Remodeling Device

INTERVENTIONS:
Device: MyoScience Tissue Remodeling Device — Percutaneous treatment with the MyoScience device

SUMMARY:
A prospective, non-randomized study to evaluate the performance of the MyoScience Tissue Remodeling Device for the treatment of glabellar lines (frown lines), lateral orbital lines (crow's feet), and frontalis lines (horizontal forehead lines).

ELIGIBILITY:
Inclusion Criteria:

* The subject must be a female 30 to 70 years of age.
* The subject must have a clinical examination prior to treatment including assessment of hyperdynamic line severity.
* The subject must have a wrinkle rating of at least "1" at rest in one or more of the following treatment areas (glabellar, lateral orbital, or frontalis).
* The subject must have signed an informed consent form.
* The subject should not have undergone any other facial cosmetic procedures at or above the level of the cheekbones within the past 6 months.
* The subject should not be participating in any other facial cosmetic research study.

Exclusion Criteria:

* The subject is on a regular regimen of prescribed or over-the-counter anticoagulants.
* The subject has an infection or skin problem at the injection site.
* The subject has a history of facial nerve palsy.
* The subject has marked facial asymmetry.
* The subject has ptosis.
* The subject has excessive dermatochalasis.
* The subject has deep dermal scarring.
* The subject has thick sebaceous skin.
* The investigator is unable to substantially lessen facial lines by physical separation.
* The subject has a history of neuromuscular disorder.
* The subject has undergone prior surgery that alters the subcutaneous anatomy of the areas being treated.
* Subjects with laxity of the canthal tendon and/or with lower lid retraction, and subjects who recruit their zygomaticus major muscle to animate their crow's feet.
* The subject has any physical or psychiatric condition that in the investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Investigators' and subjects'rating of line severity in the target areas at rest and in animation at each follow-up interval. | Up to 6 months

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Aesthetics Research Center, Redwood City, California, United States